CLINICAL TRIAL: NCT00837798
Title: Registry of AT/AF Episodes in the CRM Device Population: RATE Registry
Brief Title: RATE Registry - Registry of Atrial Tachyarrhythmia/Atrial Fibrillation (AT/AF) Episodes in the Cardiac Rhythm Management (CRM) Device Population
Acronym: RATE
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 374
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No history of AF: Patient should not have had a documented history of AF for a period of 3 months prior to enrollment.
  Interventions: Device: CRM Device

INTERVENTIONS:
Device: CRM Device — Pacemaker, ICD, or CRT device

SUMMARY:
The purpose of this registry is to produce a prospective, outcome-oriented registry to document the prevalence of AT/AF in the CRM population by using the Advanced AT/AF Diagnostics in select SJM devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient is implanted with a CRM device
* Patient has no documented history of AF (3 months prior to enrollment)
* Patient is >18 years of age
* Patient has life expectancy of >24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a CRM device
Sampling Method: Non-Probability Sample
Enrollment: 5379 (Actual)
Dates: Start 2006-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of atrial tachycardia and atrial fibrillation in a cardiac rhythm management population | 24 months

SECONDARY OUTCOMES:
Development or exacerbation of HF | 2 years
Development of AF | 2 years
AT/AF burden | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Albert Waldo, MD, Study Chair — University Hospitals Cleveland Medical Center
Locations (1):
- St Jude Medical, Sylmar, California, United States

REFERENCES:
- [Derived] Orlov MV, Olshansky B, Benditt DG, Kotler G, McIntyre T, Fujian Qu, Turkel M, Gorev M, Poghosyan H, Waldo AL. Is competitive atrial pacing a possible trigger for atrial fibrillation? Observations from the RATE registry. Heart Rhythm. 2021 Jan;18(1):3-9. doi: 10.1016/j.hrthm.2020.07.028. Epub 2020 Jul 30. PMID 32738404
- [Derived] Swiryn S, Orlov MV, Benditt DG, DiMarco JP, Lloyd-Jones DM, Karst E, Qu F, Slawsky MT, Turkel M, Waldo AL; RATE Registry Investigators. Clinical Implications of Brief Device-Detected Atrial Tachyarrhythmias in a Cardiac Rhythm Management Device Population: Results from the Registry of Atrial Tachycardia and Atrial Fibrillation Episodes. Circulation. 2016 Oct 18;134(16):1130-1140. doi: 10.1161/CIRCULATIONAHA.115.020252. PMID 27754946